CLINICAL TRIAL: NCT02198014
Title: Effectiveness of Manual Therapy and Educational Physiotherapy in the Treatment of Hemophilic Arthropathy of the Knee. A Randomized Pilot Study
Brief Title: Manual Therapy in Haemophilic Arthropathy of the Knee
Acronym: ARTHROPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, RUBÉN CUESTA-BARRIUSO, PhD, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARTHROPATHY; ARTHROPAT
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-06

CONDITIONS: Patients With Haemophilia
Keywords: Knee; Joint disease; Haemophilia; Physiotherapy modalities
MeSH Terms: conditions — Joint Diseases; Hemophilia A | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Manual Therapy group (Experimental): We employed joint traction, passive muscle stretching and isometric exercises, active resisted and proprioception exercises. The treatment in this group consisted of two sessions per week for one hour each.
  Interventions: Other: Manual Therapy
- Educational gruop (Experimental): This group received educational sessions and home exercises. The exercises are aimed at improving quadriceps strength, flexibility, range of motion and knee proprioception.
  Each educational session of 90 minute every two weeks, with exercises daily home
  Interventions: Other: Educational Physiotherapy
- Control group (No Intervention): The control group (group C) did not receive any treatment. The patients of this group were assessed by the same reviewers and under the same conditions as the subjects of the two intervention groups.

INTERVENTIONS:
Other: Manual Therapy — 5 minutes. Thermotherapy shallow to 50 cm away from the knee. 15 minutes. Joint traction, grade I-II. Fixation of distal femur with cinch and manual fixation of proximal tibia. Patient in prone position and the traction is carried out in the submaximal ranges of flexion and extension.
  10 minutes. Passive muscle stretching of quadriceps (within the limits of mobility), through compression muscle, passive muscle stretching and relaxation of muscle.
  10 minutes. Isometric and resisted exercises of quadriceps, in submaximal ranges, of flexion and extension.
  10 minutes. Proprioception exercises with unipodal support, with and without visual support, and posterior destabilization.
  10 minutes. Local cryotherapy with ice pack.
  Arms: Manual Therapy group
Other: Educational Physiotherapy — * Theory. Introduction to hemophilia: clinic and treatment; Anatomy and biomechanics of knee; Anatomy of ankle musculature; Function of muscles and haematomas treatment; Haemarthrosis, synovitis and arthropathy: clinical manifestations; Proprioception: definition and importance in hemophilia; and Physical activity and sport: risks and benefits.
  * Practice: exercises in favor of gravity; active exercises for mobility and pain management; knee proprioception exercises; isometric and isotonic exercises of quadriceps; swimming and cycling technique.
  Arms: Educational gruop

SUMMARY:
This study aims to assess the effectiveness of two Physiotherapy treatments: one with manual therapy using joint traction, passive muscle stretching, and isometric exercise, active resisted and proprioception exercises; and other treatment with educational sessions and home exercises to improve the ROM, muscle strength and proprioception in patients with haemophilia and arthropathy of the knee.

DETAILED DESCRIPTION:
Randomized trial with two treatment groups: one using joint traction, passive muscle stretching and isometric exercises, active resisted and proprioception exercises (group MT); and another with educational sessions and home exercises (group E); and a control group (group C).

The intervention was carried out during twelve weeks, performing evaluation before and after treatment, and six months of finalizing this. The treatment in MT group consisted of two sessions per week for one hour each, and the treatment in group E consisted of a session of 90 minute every two weeks, with exercises daily home. The control group (group C) did not receive any treatment. After the allocation to the groups, the composition was follows: MT group = 7; E group = 7; and control group = 7.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over the age of 18 years
* Diagnosis of haemophilia A or B
* Patients with haemophilic arthropathy in one or both knees

Exclusion Criteria:

* Patients who had a haemarthrosis of knee during intervention
* Patients with different medical diagnosis (eg, Von Willebrand's disease)
* Patients with antibodies to FVIII or FIX (inhibitors).

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in the range of movement (ROM) | Screening visit (pretreatment assessment), postreatment evaluation (12 week) and follow up assessment (6 months after treatment)
  Measurement of knee flexion and extension using a universal goniometer. Were taken as anatomical references, are indicated by Querol et al, using the reference method 0 to the mobile arm of the goniometer, as noted Norkin et al.
Changes in quadriceps muscle circumference | Screening visit (pretreatment assessment), postreatment evaluation (12 week) and follow up assessment (6 months after treatment)
  Measurement in the thigh, in two thirds of the flow distance between the anterior superior iliac spine and the joint line of the knee, using a tape measure
Changes in muscle strength of quadriceps | Screening visit (pretreatment assessment), postreatment evaluation (12 week) and follow up assessment (6 months after treatment)
  Measured by the rupture test for hemophilia patients (with a gradation of 0 to 5 points, with 0 indicating normal strength and 5 is the absence of muscle contraction).
Changes in the perception of pain | Screening visit (pretreatment assessment), postreatment evaluation (12 week) and follow up assessment (6 months after treatment)
  Using the visual analog scale, VAS, consisting of a gradation of 0 to 10 points (from no pain to worst pain imaginable).
Changes in the assessment of radiological joint deterioration | Screening visit (pretreatment assessment), postreatment evaluation (12 week) and follow up assessment (6 months after treatment)
  We use the Petterson scale which consists of 13 items (0 indicates a normal joint and joint deterioration 13 maximum).

SECONDARY OUTCOMES:
Subjects' physical characteristics | Screening visit (pretreatment assessment)
  Age of patient (years), Weight of patient (kg), Number of ankle haemarthrosis in previous year, Type of haemophilia (A or B), Severity of haemophilia (severe or moderate), Treatment (prophylaxis or on demand).
Changes in the frequency of knee hemarthrosis | Screening visit (pretreatment assessment), postreatment evaluation (12 week) and follow up assessment (6 months after treatment)
  Evaluation of knee bleeding before, during and after physiotherapy treatment. Hemarthrosis must be diagnosed clinically.

CONTACTS AND LOCATIONS:
Overall Officials: RUBEN CUESTA-BARRIUSO, PhD, Principal Investigator — Universidad Católica San Antonio
Locations (1):
- Universidad de Murcia, Murcia, Murcia, Spain

REFERENCES:
- [Derived] Cuesta-Barriuso R, Torres-Ortuno A, Nieto-Munuera J, Lopez-Pina JA. Effectiveness of an Educational Physiotherapy and Therapeutic Exercise Program in Adult Patients With Hemophilia: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 May;98(5):841-848. doi: 10.1016/j.apmr.2016.10.014. Epub 2016 Nov 16. PMID 27865846